CLINICAL TRIAL: NCT03849365
Title: Study of Erectile Dysfunction, Urinary Incontinence and Related Quality of Life After TOOKAD® Vascular Targeted Photodynamic Therapy (VTP) for Minimally Invasive Treatment of Unilateral Low Risk Prostate Cancer
Brief Title: Study of Erectile Dysfunction, Urinary Incontinence and Related QoL After TOOKAD® VTP for Low Risk Prostate Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early end of enrolment with regards to difficulty met to enrol patients
Sponsor: Steba Biotech S.A. (Other)
Collaborators: International Drug Development Institute (Other); PrimeVigilance Ltd., UK (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1802 PCM404; 2018-003228-35 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-02-21 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Low Risk Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Multiple center, single-arm, open-label, 12-month follow-up phase IV pragmatic clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOOKAD VTP (Experimental): TOOKAD is administered as part of focal VTP under general anaesthetic. TOOKAD® VTP consists of the combination of a single, 10-minute IV infusion of TOOKAD® at the dose of 3.66 mg/kg, followed by the illumination of the zone to be treated with a 753-nm laser light delivered through transperineal interstitial optical fibers at a power of 150 mW/cm and light energy of 200 J/cm applied over 22 minutes and 15 seconds.
  Interventions: Drug: TOOKAD VTP

INTERVENTIONS:
Drug: TOOKAD VTP — TOOKAD® VTP consists of the combination of a single, 10-minute IV infusion of TOOKAD® at the dose of 3.66 mg/kg, followed by the illumination of the zone to be treated with a 753-nm laser light delivered through transperineal interstitial optical fibers at a power of 150 mW/cm and light energy of 200 J/cm applied over 22 minutes and 15 seconds.

SUMMARY:
Multiple center, single-arm, open-label, 12-month follow-up phase IV pragmatic clinical trial in men with unilateral prostate cancer meeting eligibility criteria for the drug (as per the European Economic Area (EEA) Marketing Authorisation) to assess the occurrence and dynamics of the time with toxicities (urinary incontinence Grade 2 and over and/or erectile dysfunction Grade 2 and over) in patients 12 months following TOOKAD® VTP.

DETAILED DESCRIPTION:
This is a multiple center, single-arm, open-label, 12-month follow-up phase IV pragmatic clinical trial. Men with unilateral prostate cancer meeting eligibility criteria for the drug (as per the EEA Marketing Authorisation) will receive TOOKAD® VTP under general anesthesia. The primary objective is to assess the occurrence and dynamics of the time with toxicities (urinary incontinence Grade 2 and over and/or erectile dysfunction Grade 2 and over) in patients 12 months following TOOKAD® VTP. Prior to the TOOKAD® VTP, patients will undergo routine ultrasound examination in the operating room for morphometric description of the prostate and to facilitate accurate treatment guidance for the treatment with TOOKAD® VTP. Treatment will then be applied to the prostate gland as a hemi-ablation procedure designed to destroy the lobe of the prostate gland that contains the cancer. Afterwards, patients will be followed for 12 months with clinical evaluation, data collection on erectile and urinary functions at 1, 2, 3 6 and 12 months, using the Expanded Prostate Cancer Index Composite (EPIC), International Index of Erectile Function (IIEF) and International Prostate Score Symptom (IPSS) questionnaires on Quality Of Life (QOL) and Prostate Specific Antigen (PSA) testing at 3, 6 and 12 months.

The clinical follow-up of patients will follow local standard of care processes, based on recommendations in the European Summary of Product Characteristics (SmPC).

This study is a phase IV pragmatic trial using optimal dose of TOOKAD® and optimal light-energy level conditions that were determined during development and approved by the European Commission.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years of age with a life expectancy ≥ 10 years

  -.Unilateral adenocarcinoma of the prostate accurately located and confirmed as unilateral using high resolution biopsy strategies based on current best practice, such as multi- parametric MRI based strategies or template-based biopsy procedures.
* Clinical stage T1c or T2a,
* Gleason Score ≤ 6, based on high-resolution biopsy strategies
* 3 positive cancer cores with a maximum cancer core length of 5 mm in any one core or 1 -2 positive cancer cores with ≥ 50 % cancer involvement in any one core or a PSA density ≥ 0.15 ng/mL/cm3.
* PSA ≤ 10 ng/mL
* If the patient is sexually active with women who are capable of getting pregnant, he and/or his partner should use an effective form of birth control to prevent getting pregnant during a period of 90 days after the VTP procedure.
* Signed Informed Consent Form

Exclusion Criteria:

GENERAL EXCLUSION CRITERIA :

* Unwillingness to accept the treatment;
* Any previous prostatic interventions where the internal urinary sphincter may have been damaged, including trans-urethral resection of the prostate (TURP) for benign prostatic hypertrophy.
* Participation in another clinical study involving an investigational product within 1 month before study entry;
* Inability to understand the informed consent document, to give consent voluntarily or to complete the study tasks, especially inability to understand and fulfill the health-related QOL questionnaire;
* Subjects in custody and or residing in a nursing home or rehabilitation facility;
* Biopsy proven locally advanced or metastatic prostate cancer.

SURGERY AND OTHER TREATMENT-RELATED CONDITIONS OF EXCLUSION

* Any condition or history of illness or surgery that in the opinion of the investigator might affect the conduct and results of the study or pose additional risks to the subject or any medical condition that precludes the administration of a general anaesthetic or invasive procedures.
* Hypersensitivity to the active substance or to the excipient (mannitol)
* Current or prior treatment for prostate cancer.
* Patients who have been diagnosed with cholestasis.
* Current exacerbation of rectal inflammatory bowel disease.
* Anticoagulant medicinal products and those that decrease platelet aggregation (e.g. acetylsalicylic acid) should be stopped at least 10 days before the procedure with TOOKAD. Medicinal products that prevent or reduce platelet aggregation should not be started for at least 3 days after the procedure.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Cumulated time with toxicity (duration) | 12 months
  Time to onset, average duration and average time to resolution (either Erectile Dysfunction (ED) and/or Urinary Incontinence(UI)) during the 12 months following VTP of ED with severity grade 2 or over and/or UI of severity grade 2 or over, as assessed using the EPIC instrument
Cumulated time with toxicity (prevalence) | 12 months
  Prevalence at different points in time (either ED and/or UI) during the 12 months following VTP of ED with severity grade 2 or over and/or UI of severity grade 2 or over, as assessed using the EPIC instrument.
Cumulated time with toxicity (area under the curve) | 12 months
  Area under the curve with the presence of ED with severity grade 2 or over and/or UI of severity grade 2 or over, as assessed using the EPIC instrument

SECONDARY OUTCOMES:
Time with erectile dysfunction (duration) | 12 months
  Time to onset, duration, time to resolution of erectile dysfunction grade 2 or above, as assessed using the EPIC instrument
Time with erectile dysfunction (prevalence) | 12 months
  Prevalence at different points in time of erectile dysfunction grade 2 or above, as assessed using the EPIC instrument
Time with erectile dysfunction (Area under the curve) | 12 months
  Area under the curve with the presence of erectile dysfunction grade 2 or above, as assessed using the EPIC instrument
Time with urinary incontinence (duration) | 12 months
  Time to onset, duration, time to resolution of urinary Incontinence grade 2 or above, as assessed using the EPIC instrument,
Time with urinary incontinence (prevalence) | 12 months
  Prevalence at different points in time of urinary Incontinence grade 2 or above, as assessed using the EPIC instrument.
Time with urinary incontinence (Area under the curve) | 12 months
  Area under the curve with the presence of urinary Incontinence grade 2 or above, as assessed using the EPIC instrument.
Correspondence between results of EPIC and IIEF instruments | 12 months
  Average variation on urinary symptoms (UI) using the EPIC and IPSS instruments, erectile functions (ED) using the EPIC and IIEF instruments, and bowel function using the EPIC instrument, prior to treatment beginning and then at 1, 2, 3, 6 and 12 months after completing treatment: absolute scores and changes as compared to baseline (absolute difference of means and proportion change)
PSA density | 12 months
  Average changes from baseline in PSA density at month 12
Rate of Adverse Events | 12 months
  Rate of adverse events (AE) of TOOKAD® VTP treatment : all AE, important AE identified in Risk Management Plan (RMP) and suspected AE listed in RMP.
Time to resolution of Adverse events | 12 months
  Time to resolution of adverse events for each adverse event reported
Additional prostate cancer treatments | 12 months
  Rate of additional treatment as decided by local practice, such as radical therapy (surgical removal of the prostate gland, radiation treatment to the prostate gland) or other intervention therapy to the ipsilateral and/or contralateral lobe, use of hormone or chemotherapies.
Extension of prostate cancer | 12 months
  Rate of reported extension of prostate cancer based on locally decided investigations (such as clinical examination, biopsy, Magnetic resonance Imaging (MRI), other).

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Rahmène AZZOUZI, Professor, Principal Investigator — Centre Hospitalier Universitaire (CHU) ANGERS
Locations (1):
- Centre Hospitalier Universitaire (CHU), Angers, France

IPD SHARING:
Plan to Share IPD: No